CLINICAL TRIAL: NCT03804411
Title: Search for Highly Specific Predictors of Response to Different Hypoglycemic Therapy for Cardiovascular Prognosis
Brief Title: Prognostic Predictors of Response to Hypoglycemic Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other)
Responsible Party: Principal Investigator, Conrady Alexandra, Deputy General Director, Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 11/2017
Record Dates: First submitted 2018-06-08; First posted 2019-01-15 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment chosen by automated decision-making system (Experimental): Group A: type 2 diabetic patients randomized to receive antidiabetic drugs according to predictors chosen with developed automated decision-making system: subgroup 1A- addition of vildagliptin 100 mg/day, subgroup 2A - addition of sitagliptin 100 mg/day, subgroup 3A- addition of dapagliflozin 10 mg/day, subgroup 4A- addition of empagliflozin 10 mg/day, subgroup 5A- addition of liraglutide 1,2-1,8 mg/day, subgroup 6A- addition of exenatide 20 μg/day, subgroup 7A - addition of glimepiride, subgroup 8A - addition of gliclazide.
  Interventions: Drug: Automatic system guided treatment; Drug: Standard treatment
- Treatment based on standard recommendations (Experimental): Group B: type 2 diabetic patients randomized to receive antidiabetic drugs according to standard recommendations : subgroup 1B- addition of vildagliptin 100 mg/day, subgroup 2B - addition of sitagliptin 100 mg/day, subgroup 3B- addition of dapagliflozin 10 mg/day, subgroup 4B- addition of empagliflozin 10 mg/day, subgroup 5B- addition of liraglutide 1,2-1,8 mg/day, subgroup 6B- addition of exenatide 20 μg/day, subgroup 7B - addition of glimepiride, subgroup 8B - addition of gliclazide.
  Interventions: Drug: Automatic system guided treatment; Drug: Standard treatment

INTERVENTIONS:
Drug: Automatic system guided treatment — Addition of: 1A -vildagliptin 100 mg/day 2A - sitagliptin 100 mg/day, 3A- dapagliflozin 10 mg/day 4A- empagliflozin 10 mg/day 5A- liraglutide 1,2-1,8 mg/day 6A- exenatide 20 μg/day 7A - glimepiride 8A - gliclazide
Drug: Standard treatment — Addition of:
  1. B -vildagliptin 100 mg/day
  2. B - sitagliptin 100 mg/day,
  3. B- dapagliflozin 10 mg/day
  4. B- empagliflozin 10 mg/day
  5. B- liraglutide 1,2-1,8 mg/day
  6. B- exenatide 20 μg/day
  7. B - glimepiride
  8. B - gliclazide

SUMMARY:
This is a randomized controlled trial aimed to determine highly specific personified predictors of response to the therapy by different groups of hypoglycemic drugs (SGLT-2 inhibitors, DPP-4 inhibitors, GLP-1 receptor agonists, sulfonylureas) in patients with type 2 diabetes mellitus, develop an algorithm of personalized therapy based on them, design an organizational and methodological model for prevention of the cardiovascular complications, and create an automated decision-making system for therapy selection to reduce the incidence of cardiovascular events and related adverse outcomes compared to the traditional approach. This is an interventional, randomized controlled trial, open-label study.

DETAILED DESCRIPTION:
The study aims to determine highly specific personified predictors of response to the therapy by different groups of hypoglycemic drugs in patients with type 2 diabetes mellitus, to develop on their basis a mathematical model that allows to objectify the choice of therapy for each patient, and validate it in clinical practice with assessment of dynamic of cardiovascular risk markers (vascular wall condition, markers of fibrosis and inflammation, molecular-genetic markers of vascular damage, dynamic of intestinal microbiota, clinical outcomes, psychological parameters of quality of life, eating, treatment satisfaction) and pharmaco-economic component. Patients with type 2 diabetes mellitus and non-target HbA1c will be randomized to receive antidiabetic drugs (SGLT-2 inhibitors, DPP-4 inhibitors, GLP-1 receptor agonists, sulfonylureas) in open prospective study according to: 1) standard recommendations; 2) predictors chosen with automated decision-making system developed on the literature analysis. At baseline and 3, 6, 12, and 24 months into the study patients will be asked to complete the questionnaires on eating behavior, appetite, propensity to alcohol consumption, smoking, level of physical activity, general health condition, level of anxiety and depression, cognitive functions, adherence to treatment and treatment satisfaction. At baseline and 3, 6, 12, and 24 months into the study there will be physical examination and laboratory tests, including: fasting and 1.5 hours post meal glucose, glycated hemoglobin, insulin with calculation of HOMA-IR index, indicators of lipid metabolism (total cholesterol, TG, LDL, calculation of HDL and VLDL), markers of kidney function (serum creatinine with GFR calculation, urine albumin-to-creatinine ratio), biochemical parameters of therapy safety (ALT, AST, bilirubin, uric acid, fibrinogen, alkaline phosphatase, amylase 5), levels of orexigenic / anorexigenic hormones (GLP1, GIP, ghrelin, leptin, glucagon, adiponectin, C-peptide). The study will also include the evaluation of endothelial dysfunction (using EndoPAT 2000), state of the vascular wall (using the SphygmoCor), thickness of intima-media complex of carotid arteries, echocardiographic study, estimation of the global longitudinal strain (2-D Speckle-tracking echocardiographic analysis), MRI of the heart, biomarkers of inflammation (CRP level by the ultrasensitive method, adhesion molecules E-selectin and sICAM-1), markers of oxidative stress (myeloperoxidase, paraoxanase-1), markers of fibrosis (PICP, PIIINP, CITP, MMP / TIMP, TGF-β, galectin-3), markers of heart failure (NT-proBNP, sST2). The investigators will conduct immunophenotyping of circulating progenitor cells (CD45 + / CD34 + / collagen-I +) by flow cytometry, and assess molecular-genetic markers of endothelial damage (microRNA-126, microRNA-21, microRNA-27, miRNA-125 and miRoRNA-155).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female aged 17-70 years
2. Type 2 diabetes mellitus with non-target HbA1c exciding less than 1% (<1%)
3. Initiation of the treatment by SGLT- 2 inhibitors, dipeptidyl peptidase-4 inhibitors, GLP-1 analogues
4. Stable hypoglycemic therapy for 12 weeks before enrollment
5. Signed informed consent

Exclusion Criteria:

1. Type 1 diabetes mellitus
2. Recent acute coronary syndrome or acute disturbance of cerebral blood circulation (less than 2 months ago)
3. Decompensation of chronic heart failure, chronic heart failure class IV (NYHA), acute heart failure
4. Confirmed non-diabetic kidney disease (glomerulonephritis, pyelonephritis, amyloidosis)
5. Chronic kidney disease requiring hemodialysis and/or urinary albumin concentration (morning spot) >1000 mg/L
6. Regular nephrotoxic drugs intake (long-term intake of NSAIDs, aminoglycosides, sulfonamides, cyclosporine, lithium preparations)
7. Anamnesis of malignancy.
8. Diabetic foot ulcer and neuropathic osteoarthropathy
9. Anamnesis of bariatric surgery or surgical interventions on the gastrointestinal tract leading to malabsorption.
10. Treatment with drugs reducing body weight less than 3 months ago or any other drugs use that can lead to a change in body weight.
11. Liver disorders with elevation of ALT/AST exceeding three-fold the upper limit of normal
12. Immunosuppressive therapy or regular nonsteroidal anti-inflammatory drugs intake
13. Change in the dosage of thyroid hormones less than 6 weeks ago.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
HbA1c | baseline and 3, 12, and 24 months after intervention
  Change from baseline in HbA1c level (%)
Body mass index | baseline and 3, 12, and 24 months after intervention
  Change from baseline in body mass index (kg/m^2)

SECONDARY OUTCOMES:
Estimated glomerular filtration rate | baseline, 12 and 24 months after intervention
  Change from baseline in level of estimated glomerular filtration rate (ml/min/1.73 m^2)
HOMA-IR index | baseline, 6 and 12 months after intervention
  Change from baseline in level of HOMA-IR index (Homeostasis Model Assessment of Insulin Resistance) derived from the plasma insulin level (mIU/L) and plasma glucose level (mmol/L) of a participant: [(plasma insulin level) x (plasma glucose level)]/22.5, where the value of HOMA-IR index > 2.0 suggests insulin resistance
Urinary creatinine-adjusted excretion of albumin | baseline, 12 and 24 months after intervention
  Change from baseline in level of urinary creatinine-adjusted excretion of albumin in morning spot urine samples (mg/mmol)
Cardiovascular parameters of PAT and IMT | baseline, 6 and 12 months after intervention
  Change from baseline in peripheral arterial tone by using EndoPAT 2000, the thickness of intima-media complex of carotid arteries (μm)
LDL cholesterol | baseline, 6 and 12 months after intervention
  Change from baseline in level of LDL cholesterol (mmol/L)
Triglycerides | baseline, 6 and 12 months after intervention
  Change from baseline in level of triglycerides (mmol/L)
NT-proBNP | baseline, 6 and 12 months after intervention
  Change from baseline in serum level of NT-proBNP (pmol/L)
hsCRP | baseline, 6 and 12 months after intervention
  Change from baseline in serum level of hsCRP ( mg/L)
PAT | baseline, 6 and 12 months after intervention
  Change from baseline in peripheral arterial tone by using EndoPAT 2000 (Ratio is created using the post and pre occlusion values)
IMT | baseline, 6 and 12 months after intervention
  Change from baseline in the thickness of intima-media complex of carotid arteries (μm)
LV ejection fraction | baseline, 6 and 12 months after intervention
  Change from baseline in ejection fraction (%) by echocardiography
LV mass index | baseline, 6 and 12 months after intervention
  Change from baseline in LV mass index (g/m^2) by echocardiography
GLS by 2D-STE | baseline, 6 and 12 months after intervention
  Change from baseline in global longitudinal strain by 2D Speckle-tracking echocardiography (%)
Molecular-genetic markers of endothelial damage | baseline, 6 and 12 months after intervention
  Change from baseline in serum level of microRNA-126, microRNA-21, microRNA-27, miRNA-125 and miRoRNA-155 (relative units)

CONTACTS AND LOCATIONS:
Locations (1):
- Alina Babenko, Saint Petersburg, Russia